CLINICAL TRIAL: NCT00864838
Title: Effectiveness of Oral Acetazolamide, Brimonidine Tartarate, and Anterior Chamber Paracentesis for Ocular Hypertension Control After Intravitreal Bevacizumab Injection
Brief Title: Oral Acetazolamide, Brimonidine Tartarate, and Anterior Chamber Paracentesis for Ocular Hypertension Control After Intravitreal Bevacizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Apoio ao Ensino Pesquisa e Assitência do HCFMRPUSP (Unknown)
Responsible Party: Marco Antonio Bonini Filho, Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4429/2008
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Age Related Macular Degeneration; Diabetic Retinopathy
Keywords: intraocular pressure; bevacizumab; acetazolamide; brimonidine; anterior chamber paracentesis
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy | interventions — Acetazolamide; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (No Intervention): Patients submitted to 1,5 mg/0,06 ml intravitreal injection of bevacizumab and no treatment for intraocular pressure elevation
- 2 (Experimental): Acetazolamide: 250 mg of oral acetazolamide 1 hour before intravitreal bevacizumab injection
  Interventions: Drug: Acetazolamide
- 3 (Experimental): topic brimonidine tartarate: one drop of brimonidine tartarate 1 hour before intravitreal bevacizumab injection
  Interventions: Drug: Brimonidine tartarate
- 4 (Experimental): anterior chamber paracentesis: anterior chamber paracentesis immediately after intravitreal bevacizumab
  Interventions: Procedure: Anterior chamber paracentesis

INTERVENTIONS:
Drug: Acetazolamide — 250 mg 1 hour before intravitreal injection
  Other Names: Diamox
  Arms: 2
Drug: Brimonidine tartarate — 1 drop 1 hour before intravitreal injection
  Other Names: Alphagan
  Arms: 3
Procedure: Anterior chamber paracentesis — Immediately after bevacizumab injection
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the effects of anterior chamber paracentesis, brimonidine and oral acetazolamide to reduce intra-ocular pressure variations after intravitreal bevacizumab injection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of age related macular disease or diabetic retinopathy
* Able and willing to provide informed consent

Exclusion Criteria:

* History of ocular hypertension or glaucoma
* High Myopes (> 6 spherical diopters)
* High Hyperopes (> 4 spherical diopters)
* Pulmonary disease
* Renal disease
* Known allergy to any component of the study drug
* Myocardial infarction, transient ischemic attack within 4 months prior to randomization or any contraindication for bevacizumab use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (mmHg) | 1 hour and, 3 minutes before IVI. 3,10,20, 30 minutes after IVI

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Jorge, MD, Study Chair — University of Sao Paulo; Marco A Bonini-Filho, MD, Principal Investigator — University of Sao Paulo; Bianka Y Katayama, MD, Study Director — Clinic´s Hospital, Ribeirão Preto Medical School, University of São Paulo